CLINICAL TRIAL: NCT03425695
Title: Free Gingival Graft Adjunct With Low Level Laser Therapy: A Randomized Placebo- Controlled Parallel Group Study
Brief Title: Free Gingival Graft Adjunct With Low Level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Asst. Prof. Dr., Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIBU
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Wounds and Injuries; Transplants; Gingival Recession, Localized; Low-Level Light Therapy
Keywords: Free gingival graft, Low level laser therapy, Shrinkage
MeSH Terms: conditions — Wounds and Injuries; Gingival Recession | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Free Gingival Graft (FGG) + Low Level Laser Therapy (LLLT) + Clinical Examination
  The test group received LLLT with a diode laser (CheseeTM Diode Laser, Wuhan, China ) at the FGG sites with a wavelength of 810 nm and output power of 0.1 W, for 60 s, with an energy density of 6 J/cm2 in the continuous wave mode (spot size:0.5 cm). The laser beam was directed perpendicularly toward the tissue in the noncontact mode. The laser was irradiated at the recipient sites immediately after surgery and 1, 3, 7, and 14 days later.
  Interventions: Device: CheseeTM Diode Laser; Other: Clinical examination
- Control group (Placebo Comparator): Free Gingival Graft (FGG)+Placebo Low Level Laser Therapy (PLLLT) + Clinical Examination
  The control group received PLLLT with a diode laser (CheseeTM Diode Laser, Wuhan, China ) same as test group without pushing the start button
  Interventions: Device: CheseeTM Diode Laser; Other: Clinical examination

INTERVENTIONS:
Device: CheseeTM Diode Laser — low level laser therapy was utilized adjunct with free gingival graft.
Other: Clinical examination — The shrinkage of the graft area was calculated according to the differences between the graft area at baseline, 1st, 3rd, and 6th months.
  Epithelization was determined via bubbling test by using 3% hydrogen peroxide (H2O2) at 7, 14, 21, and 28 days after surgery.

SUMMARY:
The present placebo-controlled parallel design clinical study was planned to determine the effect of low level laser therapy on clinical periodontal conditions and dimensions of free gingival graft as well as postoperative pain levels in the surgical area.

DETAILED DESCRIPTION:
Background: Shrinkage of the free gingival graft (FGG) and patient's discomfort during healing period are important concerns. Therefore, this study aimed to evaluate the effect of low level laser therapy (LLLT) in terms of enhancing wound healing, reducing graft shrinkage and postoperative pain.

Methods: Thirty patients were randomly assigned to receive either FGG+ LLLT (test, n = 15) or FGG + placebo LLLT (control, n = 15). In the test group, a diode laser (aluminum-gallium-arsenide, 810 nm, 0.1 W, continuous mode, time of irradiation:60 s, energy density: 6 J/cm2, spot size:0.5 cm) was applied immediately after the FGG surgery and 1,3,7, and 14 days later. The control group received the same sequence of irradiation with the laser-off. Comparison of the graft surface areas between groups at 1st, 3rd and 6th months were made with an image-analyzing software. Complete wound epithelization, visual analogue scale (VAS) pain score of recipient site and the number of analgesic used were evaluated after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients presenting Class I or II Miller gingival recession on vital incisors in the mandibular anterior region with no caries or restoration
* The included teeth had also keratinized gingiva <2 mm; PI and GI<1.
* The patients had to be systemically healthy and non-smokers.

Exclusion Criteria:

* Patients presenting active periodontal disease and probing depth >3 mm; taking medications that would interfere with the wound-healing process or that contraindicate the surgical procedure;
* Pregnant or lactating women;
* Patients who underwent periodontal surgery in the study area;
* Patients with orthodontic therapy in progress were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Graft shrinkage | 1-, 3-, and 6-months after FGG surgery
  The shrinkage of the graft area was calculated according to the differences between the graft area at baseline, 1st, 3rd, and 6th months.

SECONDARY OUTCOMES:
Epithelization | 7, 14, 21, and 28 days after FGG surgery
  Epithelization was determined via bubbling test by using 3% hydrogen peroxide (H2O2). This test was carried out at 7, 14, 21, and 28 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: AIBU Faculty of Dentistry, Study Chair — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: Undecided